CLINICAL TRIAL: NCT04669197
Title: A Phase II Study of Paclitaxel Protein Bound + Gemcitabine + Cisplatin+ Hydroxychlororoquine as Preoperative Treatment in Patients With Untreated Resectable, Borderline Resectable and Locally Advanced Adenocarcinoma of the Pancreas
Brief Title: Study of Paclitaxel Protein Bound + Gemcitabine + Cisplatin + Hydrochloroquine as Treatment in Untreated Pancreas Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCQ NABPLAGEM-NEO 2020
Record Dates: First submitted 2020-12-01; First posted 2020-12-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Untreated Resectable Pancreatic Adenocarcinoma; Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Adenocarcinoma
MeSH Terms: interventions — Taxes; Gemcitabine; Cisplatin; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): Paclitaxel Protein Bound + Gemcitabine + Cisplatin + Hydrochloroquine
  Interventions: Drug: Paclitaxel protein bound; Drug: Gemcitabine; Drug: Cisplatin; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Paclitaxel protein bound — combination therapy
Drug: Gemcitabine — combination therapy
Drug: Cisplatin — combination therapy
Drug: Hydroxychloroquine — combination therapy

SUMMARY:
To evaluate the normalization rate of CA 19-9 of individuals with non-metastatic pancreas cancer following up to 6 months of neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically confirmed resectable, borderline resectable, or locally advanced (unresectable) PDAC (based upon Tempero et al 2016)
* Age ≥ 18 years.
* If a female patient is of child-bearing potential, she must have a negative serum pregnancy test (≥β-hCG) documented within 72 hours of the first administration of study drug
* If sexually active, the patient and partner must agree to use contraception considered adequate and appropriate by the Investigator
* Patient must have received no prior chemotherapy or radiation therapy for PDAC
* Patients must have normal organ and marrow function
* Patient has acceptable coagulation status as indicated by an INR ≤ 1.5 x ULN. Patients on anticoagulation can be included at the discretion of the investigator.
* Karnofsky Performance Status (KPS) of ≥70%.
* Have an elevated CA 19-9 (>2X ULN) in the context of normal bilirubin

Exclusion Criteria:

* Patient will be excluded from this study if any of the following criteria apply: Evidence of metastatic disease. No metastatic disease defined as any one or more of the following; Suspicious lymphadenopathy outside of the standard surgical field (i.e. aortocaval nodes, distant abdominal nodes) or Radiographic evidence for metastatic disease in distant organs, peritoneum, or ascites
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Has undergone major surgery, other than diagnostic surgery (i.e.--surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
* History of allergy or hypersensitivity to the study drugs.
* Serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
* Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
* Patient is unwilling or unable to comply with study procedures.
* Patient is enrolled in an industry sponsored clinical trial involving treatment with investigational therapy. Patients enrolled in HonorHealth sponsored research studies may be eligible to participate as long as their participation in the other research studies does not confound the data collected for this study.
* Patient with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
* Use of non-FDA approved cannabinoids are prohibited. Total daily usage of up to 40 mg per day of marinol is acceptable.

Exclusion Criteria for Hydroxychloroquine Expansion Cohort only:

* Prolonged QTcF > 450 ms for men and > 470 ms for women at Screening. Electrolyte imbalances (e.g. hypokalemia/hypomagnesemia/hypocalcemia) must be corrected prior to first dose of hydroxychloroquine.
* Known second or third degree atrioventricular block.
* Patient is taking a concomitant medication that has "known" risk of QT prolongation or torsdades de pointe.
* Patient has pre-existing retinopathy.
* Patient has known hypersensitivity to hydroxychloroquine or other 4-aminoquinoline compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Normalization Rate of CA 19-9 | 6 months
  Evaluate the normalization rate of CA 19-9 of individuals with non-metastatic pancreas cancer following up to 6 months of neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Resectability Rate | 6 months to 2 years
  Assess the resectability rate following neoadjuvant chemotherapy
Survival Rate | 2 years
  Assess the 2 year survival from date of study entry
Response Rate | 6 months to 2 years
  Assess the pathologic complete response rate and radiologic response rate
Incidence of Treatment-Emergent Adverse Events | 6 months to 2 years
  Assess the Grade 3 or Grade 4 related adverse events as assessed by CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided